CLINICAL TRIAL: NCT04228549
Title: My Peripheral Arterial Disease Management (MyPADMGT) Support of Out-Patients With Peripheral Arterial Disease
Brief Title: MyPADMGT Support of Out-Patients With Peripheral Arterial Disease
Acronym: Final_PADHSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Outpatient clinic site unable to provide required recruits due to COVID 19 virus. Terminated June 30 2022. Actual enrolment 126. This information entered August 24, 2022.
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 8108
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Usual care
- MyPADMGT (Experimental): Online access to system, with ability to record and study progress with social interaction, diet, physical activity, smoking cessation, blood glucose, blood pressure and weight. Also access to educational content, journal recording, communication to others, setting target levels, contact support as needed.
  Interventions: Device: MyPADMGT
- MyPADMGT + Nudging (Experimental): Online access to system, with ability to record and study progress with social interaction, diet, physical activity, smoking cessation, blood glucose, blood pressure and weight. Also access to educational content, journal recording, communication to others, setting target levels, contact support as needed. In addition, nudging support available to help patients make better choices and decisions.
  Interventions: Device: MyPADMGT + Nudging

INTERVENTIONS:
Device: MyPADMGT — Online tracking and feedback to help patients adopt healthy lifestyles
  Arms: MyPADMGT
Device: MyPADMGT + Nudging — Online tracking and feedback to help patients adopt healthy lifestyles plus nudging support to assist in making decisions
  Arms: MyPADMGT + Nudging

SUMMARY:
The investigators have developed an online program to help people with peripheral arterial disease (PAD) in their extremities to better self-manage their condition. Some earlier testing has been done and the investigators now wish to try this system with participants who have this blood vessel disease as well as high blood pressure. Investigators are hoping to help these participants to achieve healthier lifestyles and improve their quality of life through education, monitoring and continuing support. A similar online desk-top version with over 30 participants has been tested at St. Michael's Hospital in Toronto. The investigators propose to test this newer mobile system with 210 outpatient participants from Hamilton General Hospital. Data collected will be analyzed following the (12 months for each participant) study, along with data recorded during clinical visits at baseline and twelve months for each participant. The objective is to evaluate changes to participant health and determine whether the health self-management process has been successful in improving participant lifestyles and quality of life, when compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients with Peripheral Arterial Disease (Ankle Brachial Index < 0.90)
* Attending the Hamilton General Hospital Outpatient Vascular Clinic
* May be living alone or with one or more caregivers
* Must have Internet access.

Exclusion Criteria:

* Age < 18 years
* Not diagnosed with PAD
* Unable to communicate in English
* Unwilling to participate
* Patients with dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 1 Year
  Change in systolic blood pressure measured in clinic by blood pressure cuff
EQ-5D-5L Quality of Life Visual Result | 1 Year
  Change in QoL Visual Result measured by questionnaire. Min = 0, Max = 100. Higher outcome scores are better

SECONDARY OUTCOMES:
Ankle Brachial Index | 1 year
  Change in Ankle Brachial Index as measured in the clinic. Higher outcome scores are better
Body Weight | 1 year
  Change in Body Mass Index towards normal healthy range. Adult healthy minimum is 18.5 and healthy maximum is 24.9
Social Isolation | 1 year
  Change in Friendship Scale as measured by Hawthorne Friendship Scale Questionnaire. Min. = 0; Max. = 24. Higher outcome scores are better
Smoking Cessation | 1 year
  Smoking Cessation by Smokers as self-reported by Smokers. More Cessations is better

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stacey, MD, Principal Investigator — McMaster University
Locations (1):
- General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No